CLINICAL TRIAL: NCT01342939
Title: Postprandial Secretion of of Incretin Hormones and Incretin Effect in Patients With Maturity-onset Diabetes of the Young (MODY)
Brief Title: Pathophysiological Implications of the Incretin Hormones in Maturity Onset of Diabetes of the Young (MODY)
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other); Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Signe H Østoft, MD, MD, University Hospital, Gentofte, Copenhagen
Other Study IDs: MODY-INK; H-1-2010-130 (Registry Identifier: The Danish National Committee on Biomedical Research Ethics)
Record Dates: First submitted 2011-04-13; First posted 2011-04-27 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Maturity-onset Diabetes of the Young
Keywords: Monogenetic diabetes; Diabetes mellitus
MeSH Terms: conditions — Mason-Type Diabetes; Diabetes Mellitus | interventions — Glucose Tolerance Test; Sitagliptin Phosphate

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Buffy coat
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MODY2: Also called GCK (glucokinase) MODY. They have a specific mutation in the GCK gene.
  Interventions: Other: Oral Glucose Tolerance Test (OGTT); Other: iso glycaemic intravenous (iv) glucose infusion (IIGI); Dietary Supplement: Meal test; Other: Incretin effect on sulphonyl urea treatment
- MODY3: Also called HNF1 alfa MODY. They have a specific mutation in the HNF1 alfa gene.
  Interventions: Other: Oral Glucose Tolerance Test (OGTT); Other: iso glycaemic intravenous (iv) glucose infusion (IIGI); Dietary Supplement: Meal test; Other: Incretin effect on sulphonyl urea treatment
- Healthy control subjects
  Interventions: Other: Oral Glucose Tolerance Test (OGTT); Other: iso glycaemic intravenous (iv) glucose infusion (IIGI); Dietary Supplement: Meal test; Other: Sitagliptin

INTERVENTIONS:
Other: Oral Glucose Tolerance Test (OGTT) — 50g waterfree glucose dissolved in 300ml water consumed over 5 min.
  Other Names: Waterfree glucose, The Pharmacy of the capital region
Other: iso glycaemic intravenous (iv) glucose infusion (IIGI) — 20% glucose
  Other Names: Glucose infusion, 20%
Dietary Supplement: Meal test — Energy drink, 350ml (525 kcal: 65 g carbohydrates, 20 g fat and 21 g protein)
  Other Names: Nutridrink with cocoa taste (Nutricia, Allerød, Denmark)
Other: Sitagliptin — Healthy control subject are given an acute dosage of 100mg the evening before the experimental day, and the same morning in order to increase levels of endogen incretin hormones
  Other Names: Januvia, 100mg
  Groups: Healthy control subjects
Other: Incretin effect on sulphonyl urea treatment — Subject with MODY who are treated with sulphonyl urea are investigated without medication break prior to examination.
  Groups: MODY2; MODY3

SUMMARY:
The purpose of this study is to describe the incretin effect and postprandial incretin response in patients with MODY2 and MODY3 and a group of matched healthy subjects. In sulphonyl urea treated subjects the purpose is also to compare the incretin effect with and without treatment. In healthy subjects the purpose is also to investigate the incretin effect under increased levels of endogen incretin hormones.

DETAILED DESCRIPTION:
Comparison of of insulin secretion (AUC) during the experimental days. Furthermore a comparison of GIP, GLP1 and glucagon responses as well as plasma glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians above 18 years
* BMI > 19 kg/m2
* Negative pancreatic beta cell- and glutamate decarboxylase-65(GAD65)- autoantibodies
* Normal haemoglobin
* Normal bloodpressure
* Informed concent

Exclusion Criteria:

* Known liver disease or affected liver enzymes (ALAT/ASAT >2 x upper normal limit)
* Nephropathy (see creatinine> 130 μM and / or albuminuria)
* Treatment with medications that cannot be discontinued for 12 hours
* Any condition that the investigators feel would interfere with trial participation
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Genetically well-charaterized MODY2 and MODY3 patients at Hagedorn Research Institute/Steno Diabetes Center
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incretin effect | Within 1 year
  The difference in insulin responses, as assessed by the area under curve (AUC) for plasma insulin and C-peptide concentrations, during the two different glucose stimuli: OGTT and isoglycemic iv glucose infusion aswell as after a test meal in MODY-patients compared to healthy control subjects.

SECONDARY OUTCOMES:
Plasma GLP1 response | Within 1 year
  Comparing GLP1 responses of the different experimental days, compared to healthy control subjects.
Plasma GIP response | Within 1 year
  Comparing GIP responses of the different experimental days, compared to healthy control subjects.
Plasma glucagon response | Within 1 year
  Comparing glucagon responses of the different experimental days, compared to healthy control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Signe H Østoft, MD, phd stud, Principal Investigator — Diabetes Research Division, University Hospital Gentofte, Denmark
Locations (1):
- Diabetes Research Division, Gentofte University Hospital, Niels Andersens vej 65, opgang 40, 2., Hellerup, Denmark

REFERENCES:
- [Derived] Ostoft SH, Bagger JI, Hansen T, Hartmann B, Pedersen O, Holst JJ, Knop FK, Vilsboll T. Postprandial incretin and islet hormone responses and dipeptidyl-peptidase 4 enzymatic activity in patients with maturity onset diabetes of the young. Eur J Endocrinol. 2015 Aug;173(2):205-15. doi: 10.1530/EJE-15-0070. Epub 2015 May 7. PMID 25953829